CLINICAL TRIAL: NCT05735561
Title: Association Between the Direction of Proximal Humerus Fracture Dislocation and Risk of Avascular Necrosis Following Open Reduction Internal Fixation - An Observational, Cohort Study
Brief Title: Proximal Humerus Fracture Dislocation Direction and Avascular Necrosis
Acronym: PHF-D
Status: Completed | Type: Observational
Sponsor: Fraser Orthopaedic Research Society (Network)
Responsible Party: Sponsor
Other Study IDs: 2023-006
Record Dates: First submitted 2023-01-27; First posted 2023-02-21 (Actual); Last update posted 2023-09-13 (Actual); Status verified 2023-09

CONDITIONS: Proximal Humeral Fracture; Dislocation; Dislocation Shoulder; Avascular Necrosis; Avascular Necrosis of Humerus
MeSH Terms: conditions — Shoulder Fractures; Joint Dislocations; Shoulder Dislocation; Osteonecrosis | interventions — X-Rays

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Proximal Humerus Fracture Anterior Dislocation: The study doesn't provide any intervention. This group is defined as having a dislocation that is anterior to the glenoid.
- Proximal Humerus Fracture Posterior Dislocation: The study doesn't provide any intervention. This group is defined as having a dislocation that is posterior to the glenoid.
  Interventions: Diagnostic Test: X-Ray
- Proximal Humerus Fracture Varus Dislocation: The study doesn't provide any intervention. This group is defined as having a dislocation that is in varus compared to the glenoid.
  Interventions: Diagnostic Test: X-Ray
- Proximal Humerus Fracture Valgus Dislocation: The study doesn't provide any intervention. This group is defined as having a dislocation that is in valgus compared to the gelnoid.
  Interventions: Diagnostic Test: X-Ray

INTERVENTIONS:
Diagnostic Test: X-Ray — Consenting participants will be asked to come into the clinic for a single visit, during this visit they will be asked to complete an x-ray to check for evidence of avascular necrosis.
  Groups: Proximal Humerus Fracture Posterior Dislocation; Proximal Humerus Fracture Valgus Dislocation; Proximal Humerus Fracture Varus Dislocation

SUMMARY:
The purpose of the study is to see if there is a connection between a proximal humerus fracture dislocation direction and the likelihood of developing avascular necrosis. Utilizing a retrospective cohort from the last ten years we hope to bring consenting patients back for a single visit to have x-rays and complete patient reported outcome measures to assess for evidence of avascular necrosis.

DETAILED DESCRIPTION:
The incidence of proximal humerus fractures continues to increase and is among one of the more common fractures seen in the adult population. Proximal humerus fracture dislocations, however, are less common. Despite the decreased prevalence, fracture dislocations have unique challenges with respect to obtaining an anatomical reduction and more frequently involve an open surgical reduction. In addition, depending on other fracture characteristics, there are various treatment options for the fracture itself. While fracture dislocations ultimately lead to increased AVN and revision surgery, further discussion surrounding the direction of dislocation and how it may influence overall outcomes has not been addressed in the previous literature. The study design utilizes a retrospective cohort from the last ten years, by asking patients who have had a previously surgically treated proximal humerus fracture dislocations to come back to the surgeon's private clinic to complete a single visit assessment. During this assessment the consenting participant will receive x-rays and complete patient reported outcome measures. In conjunction, these will be utilized to assess overall function and the existence of avascular necrosis.

ELIGIBILITY:
Inclusion Criteria:

* Patients 18 years of age or older
* Patients who underwent operative fixation of proximal humerus fracture dislocation at Royal Columbian Hospital between January 2011 and July 2021
* Willing and able to consent and complete patient reported outcome measures
* Willing and able to follow the protocol and attend a follow-up visit
* Able to read and understand English or have an interpreter available

Exclusion Criteria:

* Skeletally immature patients
* Patient with pathological fractures
* Patients who have had previous operative fixation of proximal humerus
* Patients treated non-operatively
* patients presenting outside of the study duration window
* Patients treated by a non-participating surgeon
* Deceased patients
* Patients unable to complete patient reported outcome measures
* Patients declining to come back to the clinic for updated x-rays
* Dementia
* Incarceration

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Skeletally mature patients who were surgically treated for their proximal humerus fracture dislocation between 2011 and 2021.
Sampling Method: Non-Probability Sample
Enrollment: 25 (Actual)
Dates: Start 2023-02-15 (Actual); Primary Completion 2023-07-31 (Actual); Study Completion 2023-08-31 (Actual)

PRIMARY OUTCOMES:
Rates of Avascular Necrosis | At least 2 years post fracture fixation
  The presence and advancement of avascular necrosis (as classified by the Cruess Classification System) and as assessed on radiographs.
Direction of the Humeral Fracture Dislocation | At least 2 years post fracture fixation
  As characterized by the direction of the humeral head in relation to the glenoid, based on AP, Lateral, or Axillary x-ray views.

SECONDARY OUTCOMES:
DASH (functional outcome) | At least 2 years post fracture fixation
  Asking participants to complete the Disabilities of the Arm, Shoulder, and Hand outcome measure as a way of assessing function.
Constant Score (functional outcome) | At least 2 years post fracture fixation
  Asking participants to complete the Constant Score patient reported outcome measure as a way of assessing participant function.

CONTACTS AND LOCATIONS:
Overall Officials: Farhad Moola, MD, Principal Investigator — FHA Orthopaedic Surgeon
Locations (1):
- Royal Columbian Hospital/Fraser Health Authority, New Westminster, British Columbia, Canada

IPD SHARING:
Plan to Share IPD: No
There is currently no plan to share individual participant data with other researchers, results will of course be shared. However, the hope is that the study might indicate a need for a high powered prospective clinical trial to be completed.

REFERENCES:
- [Background] Schumaier A, Grawe B. Proximal Humerus Fractures: Evaluation and Management in the Elderly Patient. Geriatr Orthop Surg Rehabil. 2018 Jan 25;9:2151458517750516. doi: 10.1177/2151458517750516. eCollection 2018. PMID 29399372
- [Background] Greiner S, Kaab MJ, Haas NP, Bail HJ. Humeral head necrosis rate at mid-term follow-up after open reduction and angular stable plate fixation for proximal humeral fractures. Injury. 2009 Feb;40(2):186-91. doi: 10.1016/j.injury.2008.05.030. Epub 2008 Dec 18. PMID 19100544
- [Background] Hertel R, Hempfing A, Stiehler M, Leunig M. Predictors of humeral head ischemia after intracapsular fracture of the proximal humerus. J Shoulder Elbow Surg. 2004 Jul-Aug;13(4):427-33. doi: 10.1016/j.jse.2004.01.034. PMID 15220884
- [Background] Boesmueller S, Wech M, Gregori M, Domaszewski F, Bukaty A, Fialka C, Albrecht C. Risk factors for humeral head necrosis and non-union after plating in proximal humeral fractures. Injury. 2016 Feb;47(2):350-5. doi: 10.1016/j.injury.2015.10.001. Epub 2015 Oct 22. PMID 26706457
- [Background] Miltenberg B, Masood R, Katsiaunis A, Moverman MA, Puzzitiello RN, Pagani NR, Menendez ME, Salzler MJ, Drager J. Fracture dislocations of the proximal humerus treated with open reduction and internal fixation: a systematic review. J Shoulder Elbow Surg. 2022 Oct;31(10):e480-e489. doi: 10.1016/j.jse.2022.04.018. Epub 2022 May 20. PMID 35605847
- [Background] Cruess RL, Blennerhassett J, MacDonald FR, MacLean LD, Dossetor J. Aseptic necrosis following renal transplantation. J Bone Joint Surg Am. 1968 Dec;50(8):1577-90. No abstract available. PMID 4881164

DOCUMENTS (2):
  • Study Protocol (2023-01-09): https://cdn.clinicaltrials.gov/large-docs/61/NCT05735561/Prot_000.pdf
  • Informed Consent Form (2023-01-24): https://cdn.clinicaltrials.gov/large-docs/61/NCT05735561/ICF_001.pdf